CLINICAL TRIAL: NCT06603363
Title: Changes in Plaque Characteristics After Short-term Statin Therapy as Assessed With Coronary CT
Acronym: INTENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Maurovich-Horvat Pál (Other)
Collaborators: National Research, Development and Innovation Office, Hungary (Unknown); HeartFlow, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Prof. Maurovich-Horvat Pál, Head of Clinic for Medical Imaging, Semmelweis University
Organization: Semmelweis University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BM/17433-1/2024; 2025-521367-12-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease; Atherosclerotic Plaque; Coronary Computed Tomography Angiography; Statin Therapy; Multidetector Computed Tomography; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Vascular Diseases; Hyperlipidemia
Keywords: coronary artery disease; stable chest pain; intermediate pretest probability; explanatory randomised controlled trial; coronary computed tomography angiography; photon-counting detector CT; atherosclerotic plaque; statin therapy
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Vascular Diseases; Hyperlipidemias | interventions — Rosuvastatin Calcium; Hematologic Tests; Clinical Laboratory Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensified Statin Arm (Experimental): Participants will receive one capsule (40 mg of rosuvastatin), taken once daily for 3 months, orally with or without food. After the 3-month visit, the dose will be reduced to a dose per standard of care.
  Interventions: Drug: Rosuvastatin 40mg; Diagnostic Test: Coronary Computed Tomography Angiography (Coronary CTA); Diagnostic Test: Blood test
- Placebo Arm (Placebo Comparator): Participants will receive one capsule (a placebo for rosuvastatin), taken once daily for 3 months, orally with or without food. After the 3-month visit standard rosuvastatin therapy will be initiated.
  Interventions: Drug: Placebo; Diagnostic Test: Coronary Computed Tomography Angiography (Coronary CTA); Diagnostic Test: Blood test

INTERVENTIONS:
Drug: Rosuvastatin 40mg — Participants will receive 40 mg of rosuvastatin once a day for 3 months. After the 3-month visit, the dose will be reduced to a dose per standard of care.
  Other Names: Intensified Statin Therapy
  Arms: Intensified Statin Arm
Drug: Placebo — Participants will receive a placebo for rosuvastatin once a day for 3 months. After the 3-month visit, standard rosuvastatin will be initiated.
  Arms: Placebo Arm
Diagnostic Test: Coronary Computed Tomography Angiography (Coronary CTA) — Computed Tomography Angiography including coronary calcium scoring and coronary computed tomography angiography at baseline, 3-month, and 24-month visits with a PCD-CT scanner.
  Other Names: Coronary CTA
Diagnostic Test: Blood test — Blood test at baseline, 3-month, and 24-month visits.
  Other Names: Laboratory test

SUMMARY:
INTENSE Trial is a prospective, double-blind, randomized, placebo-controlled, single-center study with two arms (40 mg intensified statin therapy vs matching placebo for rosuvastatin) among statin-naive patients referred to coronary CT angiography due to stable chest pain, followed for 24 months by using a photon-counting detector CT (PCD-CT).

INTENSE Trial aims 1) to assess the effect of short-term intensified statin therapy on coronary anatomy and physiology using PCD-CT and 2) to determine the impact of short-term, intensified statin therapy on coronary plaque morphology and hemodynamics to identify statin responder and non-responder patients in addition to testing the hypothesis of "plaque memory" after the 24-month follow-up period.

DETAILED DESCRIPTION:
The extent to which short-term intensified statin treatment may modulate plaque lipid content, alter plaque structure, and change flow physiology as assessed by non-invasive imaging remains unknown. Furthermore, no data is available regarding the effects of short-term intensified statin therapy on coronary plaques as assessed by Photon-Counting Detector CT (PCD-CT). In addition, no data is available regarding the long-term effects of short, intensified statin therapy on plaque morphology (i.e., plaque memory). Therefore, in this randomized, controlled, prospective, double-blind, single-center clinical trial, we aimed 1) to assess the effect of short-term intensified statin therapy on coronary anatomy and physiology using PCD-CT and 2) to assess the effect of short, intensified statin treatment on long term changes in plaque characteristics. In other words, to test our "plaque memory" hypothesis. Our analyses include a detailed evaluation of plaques by combining anatomic (quantitative and qualitative plaque assessment, radiomics) and hemodynamic (Fractional Flow Reserve-CT, FFR-CT) information.

In this randomized, controlled, prospective double-blinded single-center clinical trial, we aim to enroll statin naive patients (patients with no previous or current statin treatment) who underwent PCD-CT (NAEOTOM Alpha, Siemens Healthineers, Erlangen, Germany) exam due to stable chest pain and suspected coronary artery disease (CAD) at the Medical Imaging Centre of Semmelweis University, Budapest, Hungary. Coronary CT Angiography (Coronary CTA) examinations will be performed in accordance with the current guidelines of the Society of Cardiovascular Computed Tomography.

We will enroll patients aged 30-65 years, with at least one partially calcified or non-calcified plaque and with negative FFR-CT (FFR-CT>0.75 distal to stenosis).

Patients with contraindications to coronary CTA and patients post-revascularisation will be excluded from the study. Additional exclusion criteria: patients receiving lipid-lowering therapy before coronary CTA exam; alanine aminotransferase (ALT) levels >3× upper limit of normal (ULN); unexplained serum creatine kinase (CK) level >3× ULN; serum creatinine >2 mg/dL (177 umol/l), elevated low-density lipoprotein (LDL) level >5 mmol/L.

Patients will be randomized into 'high-dose statin' and 'placebo' groups, considering the age and sex of the patients to achieve equal representation of age groups and genders in both arms. Based on the sample size calculation, 70-70 patients must be randomized into each group. For those who will be randomized to the 'high-dose statin' group, 40 mg rosuvastatin therapy will be initiated. For those who will be randomized to the 'placebo' group, a placebo therapy will be started with medications that look the same as 40 mg rosuvastatin pills.

All the included patients will undergo repeated coronary CTA at 3 months and 24 months after the baseline CT. After the 3-month coronary CTA control, rosuvastatin dose per standard of care will be initiated. The 3-month and 24-month control coronary CTA evaluations will be the same as the baseline CT scans. All coronary CTA exams will be performed using a low radiation dose protocol utilizing the advanced imaging capabilities of PCD-CT.

All the included patients will undergo repeated coronary CTA at 3 months and 24 months after the baseline CT with a standardized acquisition protocol.

Proposed scan parameters for all patients are as follows: tube voltage = 120 kVp (due to improved spectral data), automatic tube current modulation with image quality level (IQ-level) = 80, detector configuration = 144 mm × 0.4 mm, rotation time = 0.25 s. All coronary CTA exams will be performed by using a low radiation dose protocol utilizing the advanced imaging capabilities of PCD-CT.

Patients may receive intravenous or oral beta blockers if their heart rate (HR) is > 65 beats/minute before the examination. All patients will receive a nitroglycerine transdermal patch before CTA scanning if systolic blood pressure is > 100 Hgmm. Prospectively triggered acquisition mode is preferred in case of regular HR > 70 beats/min, and helical scan mode if HR is irregular. Images will be acquired in diastole (65-85% of the R-R interval) or systole (200-400 ms), depending on the HR (< or > 75 beats/minute). A four-phasic contrast injection protocol with 70-80 mL contrast agent at a flow rate of 4.5-5.0 mL/s is recommended.

Special attention will be given to ensure that the baseline CT scan parameters are consistent with the follow-up scans for each patient. Images and coronary segments with severe motion, breathing, beam-hardening, or misalignment artifacts will be excluded from the analysis. Coronary segments matched to the segment with artifacts will also be excluded in all scans.

The primary endpoint will be evaluated at 3 months, while "plaque memory" will be assessed at 24 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for coronary computed tomography angiography (CTA)
* females aged 45-75 years and males aged 40-75 years
* presence of at least mild coronary atherosclerosis (luminal stenosis >25%, with at least one partially calcified or non-calcified plaque)
* statin-naive patients
* ability to understand and provide written informed consent
* FFR-CT value ≥0.75, indicating the absence of hemodynamically significant stenosis

Exclusion Criteria:

* contraindications to coronary CTA
* current or prior treatment with statins or other lipid-lowering agents (e.g., ezetimibe)
* age below 45 years in females or below 40 years in males
* age above 75 years in both sexes
* pregnancy or breastfeeding
* type 1 or type 2 diabetes mellitus
* history of coronary stent implantation or coronary artery bypass grafting
* history of myocardial infarction
* ≥70% luminal stenosis in the proximal left anterior descending artery (LAD), or ≥50% stenosis in the left main (LM) coronary artery
* FFR-CT value <0.75 in any coronary artery
* elevated serum alanine aminotransferase (ALT) levels (>3× the upper limit of normal)
* elevated serum creatine kinase (CK) levels (>3× the upper limit of normal)
* LDL cholesterol level >5 mmol/L
* renal failure or significantly impaired renal function (eGFR <30 mL/min/1.73 m²)
* ongoing oncological treatment
* active liver disease
* known hypersensitivity to any excipients of the investigational product
* concomitant treatment with the combination of sofosbuvir/velpatasvir/voxilaprevir
* concomitant treatment with cyclosporine
* women of childbearing potential not using adequate contraception
* presence of myopathy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in non-calcified plaque volume during a 3-month follow-up period. | 12 weeks
  Expressed as absolute change and as a percentage of baseline.

SECONDARY OUTCOMES:
Change in total plaque volume at 3-month follow-up period. | 12 weeks
  Expressed as change in total plaque volume (mm3) at 3-month follow-up.
Change in low attenuation non-calcified plaque volume during a 3-month follow-up period. | 12 weeks
  Expressed as absolute change and as a percentage of baseline.
Change in low attenuation non-calcified plaque volume during a 24-month follow-up period. | 24 months
  Expressed as absolute change and as a percentage of baseline.
Change in total plaque volume during a 24-month follow-up period. | 24 months
  Expressed as absolute change and as a percentage of baseline.
Change in total plaque volume between 3- and 24-month follow-up period. | 21 months
  Expressed as absolute change and as a percentage of 3-month follow up.
Change in non-calcified plaque volume between 3- and 24-month follow-up period. | 21 months
  Expressed as absolute change in non-calcified plaque volume (mm3) of 3-month follow up.
Change in non-calcified plaque volume during a 24-month follow-up period. | 24 months
  Expressed as absolute change and as a percentage of baseline.
Change in plaque composition during a 3-month follow-up period. | 12 weeks
  Plaque components are defined based on the following Hounsfield Unit (HU) threshold ranges: Low-attenuation plaque: - 100 to 30 HU; Non-calcified plaque: 30 to 350 HU; Calcified plaque: above 350 HU. Plaque components will be combined to report volumetric change in mm3.
Change in plaque composition during a 24-month follow-up period. | 24 months
  Plaque components are defined based on the following Hounsfield Unit (HU) threshold ranges: Low-attenuation plaque: - 100 to 30 HU; Non-calcified plaque: 30 to 350 HU; Calcified plaque: above 350 HU. Plaque components will be combined to report volumetric change in mm3.
Change in per-vessel fractional flow reserve [FFRCT] during a 3-month follow-up period. | 12 weeks
  CT-derived fractional flow reserve [FFRCT] will be calculated using computational fluid dynamics with off-site supercomputers. FFRCT values defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Change in per-vessel fractional flow reserve [FFRCT] during a 24-month follow-up period. | 24 months
  CT-derived fractional flow reserve [FFRCT] will be calculated using computational fluid dynamics with off-site supercomputers. FFRCT values defined as follows: greater than 0.8 is normal, 0.76-0.8 is borderline, and 0.75 or less is abnormal.
Change in the prevalence of high-risk plaque features during a 3-month follow-up period. | 12 weeks
  Low attenuation plaque, positive remodeling, napkin-ring sign, spotty calcification, minimal luminal area or plaque burden ≥70% will be combined to report high risk plaque features in numbers.
Change in the prevalence of high-risk plaque features during a 24-month follow-up period. | 24 months
  Low attenuation plaque, positive remodeling, napkin-ring sign, spotty calcification, minimal luminal area or plaque burden ≥70% will be combined to report high risk plaque features in numbers.
Change in radiomic features during a 3-month follow-up period. | 12 weeks
  Radiomic features are defined as first-order metrics (describing the distribution of HU values); gray-level co-occurrence matrix (GLCM) textural parameters (describing how often voxels of a similar value occur next to each other) and geometric parameters (describing spatial characteristics such as shape, size, or volume).Radiomic features will be calculated for each segmentation mask (defined as plaque).
Change in radiomic features during a 24-month follow-up period. | 24 months
  Radiomic features are defined as first-order metrics (describing the distribution of HU values); gray-level co-occurrence matrix (GLCM) textural parameters (describing how often voxels of a similar value occur next to each other) and geometric parameters (describing spatial characteristics such as shape, size, or volume).
Prevalence of major adverse cardiac event | From inclusion up to a maximum follow-up period of 4 years
  Composite endpoint: major adverse cardiovascular event (MACE) defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, stroke. Prevalence will be calculated as the percentage of patients who suffered MACE.
Prevalence of clinical adverse event | From inclusion up to a maximum follow-up period of 4 years
  Composite endpoint: defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, stroke, unstable angina, or heart failure admission. Prevalence will be calculated as the percentage of patients who suffered one the above listed.
Reproducibility of quantitative plaque assessment | 12 weeks
  Retrospective analysis of the reproducibility of quantitative plaque assessment in patients assigned to the placebo arm at the 3-month follow-up period. Plaque components are defined based on the following Hounsfield Unit (HU) threshold ranges: Low-attenuation plaque: - 100 to 30 HU; Non-calcified plaque: 30 to 350 HU; Calcified plaque: above 350 HU. Plaque components will be combined to report volumetric change in mm3.

OTHER OUTCOMES:
Changes in blood lipid profile | Measured at baseline, at 3-month and 24-month
  Expressed as change from baseline in total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, LP(a), apoA1 and apoB levels.
Changes in inflammatory markers | Measured at baseline, at 3-month and 24-month
  Expressed as change in hs-CRP and ferritin.
Changes in markers of glucose homeostasis | Measured at baseline, at 3-month and 24-month
  Expressed as change in hemoglobin A1c.

CONTACTS AND LOCATIONS:
Overall Officials: Pál Maurovich-Horvat, Prof., Dr., Principal Investigator — Medical Imaging Centre, Budapest, Hungary; Marc Dewey, Prof., Dr., Study Chair — Charite University, Berlin, Germany; Béla Merkely, Prof., Dr., Study Chair — Heart and Vascular Centre, Budapest, Hungary
Locations (1):
- Semmelweis University, Medical Imaging Centre, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
GUIDE-IT platform (www.guide-it.org) will be used for sharing clinical and imaging data after results are published.
Time Frame: Clinical and imaging data will be available after the results have been published.
Access Criteria: Access request needs to be made directly to the PI.